CLINICAL TRIAL: NCT03991351
Title: Investigation Into the Impact of Exposure to Images of the Idealised Physique on Body Satisfaction, Dieting Intentions and Mood in Men.
Brief Title: Impact of Exposure to Images of the Idealised Physique on Body Satisfaction, Dieting Intentions and Mood in Men.
Status: Completed | Type: Observational
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Dr Graham Finlayson, Professor, University of Leeds
Other Study IDs: PSC-670
Record Dates: First submitted 2019-05-15; First posted 2019-06-19 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Body Image
Keywords: Body Image; Mood, anxiety, depression; Self-esteem; Body Dysmorphia; Men; Deit; Exercise
MeSH Terms: conditions — Anxiety Disorders; Depression; Multiple Endocrine Neoplasia Type 1; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Men aged 18-34: Participants will be males aged 18-34. Each individual will be exposed to images of men with either a muscular, skinny or overweight physique or the control images of landscapes.
  Interventions: Other: Exposure to images

INTERVENTIONS:
Other: Exposure to images — Exposure to images

SUMMARY:
Every day, people are exposed to huge amounts of media. Research has explored the impact of viewing traditional media and advertising (such as television and magazines) on how a person thinks and feels about their body (body satisfaction). However, less is known about the impact of exposure to social media on body satisfaction. It is important to consider this now, given the rise in social media use.

The rise in social media use has made it easier for people to share images of an 'ideal' body, which for men is high muscularity and low body fat. Alongside this rise in the ideal body being shared on social media, there is a rise in male eating disorders. Research has already demonstrated that showing images of the 'ideal' body decreases body satisfaction. However, there has been little research in men and this research uses media from magazines.

The present study will update research by using images taken from Instagram and by recruiting male participants. Participants will be asked to take part in an online survey (shared on social media) which measures initial mood, body satisfaction, self-esteem and diet and exercise intentions. It will then show participants images of men with different physiques (either muscular, overweight, slender or control images of landscapes). The measures will then be repeated to see if viewing the images had any impact

DETAILED DESCRIPTION:
The present study will seek to replicate findings of previous studies by exposing men to images of the idealised male physique and demonstrating increased body dissatisfaction and negative affect. However, given the rise of social media and the suggestion that social media platforms should be investigated independently, the present study aims to update literature by using images from Instagram rather than traditional forms of media. Instagram was chosen based on the suggestion that this social media platform may be the most detrimental to body image concerns because of its sole focus on photo activity and hence the elevated opportunity for social comparison. Additionally, male participants were chosen because to the author's knowledge, the experimental studies which have exposed participants to images taken from Instagram have only recruited women.

This study also builds upon previous findings that exposure impacts upon eating disorder and muscle dysmorphia symptomatology, by ensuring that the measures used to investigate these constructs are more relevant and more valid in men. This is achieved by measuring men's intentions to modify their diet and exercise regime to increase muscularity. Dieting and exercise intentions are measured, given the limitations in directly monitoring diet and exercise through diaries and according to the theory of planned behaviour, intentions strongly predicts actual behaviour. Pre and post exposure scores are used to investigate whether exposure has an impact on these outcomes.

Moderating factors such as gym use, pre-existing body and muscle dissatisfaction and social media use are controlled for in hope of demonstrating larger effect sizes. The reason for this is because the above research suggests that those using social media more often, those not attending the gym and those with pre-existing body or muscle dissatisfaction are more at risk of body dissatisfaction and other negative effects following exposure to images of the idealised physique.

This study also builds upon research which has provided evidence for the processes underlying the relationship between exposure to idealised images and body dissatisfaction. Research suggests that social comparison is a mediating factor, however this research either draws upon traditional media rather than social media to source images or the research only utilises female participants. Therefore, this study combines the use of images taken from Instagram with the recruitment of male participants. Additionally, in the hope of providing stronger evidence for underlying processes, social comparison is measured directly (instead of being inferred). Given the suggestion that people are more likely to socially compare themselves to peers rather than models or celebrities, images used in exposure did not include models or celebrities.

Finally, this study will learn from limitations of other studies by dividing their 'average' condition into two (skinny and overweight) in addition to maintaining a muscular and control group. The purpose of this is to demonstrate the role of upward and downward social comparisons to support the social comparison theory as an explanation of the effect.

The study utilises an experimental design as there is sufficient literature to generate hypotheses to be tested. Additionally, an experimental design is a robust and controlled method of capturing the acute effects of manipulating an independent variable.

The study adopts a between subjects design with four conditions. Each participant will complete one of four online questionnaires on SurveyMonkey. The four questionnaires are identical except for the images contained within them, hence the independent variable is image type. Each questionnaire will contain 15 images of either the idealised physique (muscular, lean and low body fat), overweight physique, skinny physique or landscapes (control images). These images will be selected from a pool of images by an independent panel in the target age range in the initial stage of the study.

ELIGIBILITY:
Inclusion Criteria:

* Any men aged 18-34

Exclusion Criteria:

* Females, current or historical diagnosis of eating disorders, anyone who falls outside of age limit

Ages: 18 Years to 34 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Any men aged 18-34 will be recruited. Students from the University of Leeds will make up a large proportion of the sample.
Sampling Method: Non-Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
State Body Satisfaction | Through study completion. Participants are asked to rate their current body satisfaction before they view the images (after approx 5 minutes) and are asked the same questions again immediately after they view the images (after approx 10-15 minutes)
  Visual Analogue Scale of body satisfaction. Each item is scored by participants between 0-100 (0 = not at all satisfied, 100 = very satisfied).

SECONDARY OUTCOMES:
Diet and Exercise Intentions | Participants are asked to rate their intentions to change their diet and exercise (over the next 2-3 days) before they view the images and again immediately after they view the images.
  Measures participants intentions to change their diet and exercise type/frequency. Measured using a 7 point likert scale where 1 = strongly disagree and 7 = strongly agree.

OTHER OUTCOMES:
Mood | Through study completion. Participants are asked to rate their current mood before they view the images (after approx 5 minutes) and are asked the same questions again immediately after they view the images (after approx 10-15 minutes).
  Individual Visual Analogue Scales for anxiety, depression, confidence, anger and happiness. Each item is scored by participants between 0-100 (0= not at all anxious, depressed, angry, happy, confident and 100 = very anxious, depressed, angry, confident, happy).
State Self-esteem scale (appearance subscale) | Through study completion. Participants are asked to rate how they feel in response to the questions before they view the images (after approx 5 minutes) and are asked the same questions immediately after they view the images (after approx 10-15 minutes).
  Measure of self-esteem using a 5 point likert scale ranging from 1-5 (1=not at all true, 5=extremely true)
State Appearance Comparison | Through study completion. Participants are asked to rate this measure immediately after they have viewed the images (after approx 15 minutes).
  Measure of comparison of own body to images viewed in the questionnaire. Measured using a 7 point likert scale (1=no thought about my appearance when viewing the images, 7 = a lot of thought about my appearance when viewing the images).
Trait body satisfaction | Participants rate the questions in this measure once at baseline after approx 5 minutes (before the images are presented to them)
  Measure of trait (baseline) body satisfaction. Measured on a 6 point likert scale (1=never, 6=always).

CONTACTS AND LOCATIONS:
Locations (1):
- Online, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data will not be made publicly available. Data may be made available for relevant future research upon reasonable request to the research supervisor.

REFERENCES:
- [Background] Blond A. Impacts of exposure to images of ideal bodies on male body dissatisfaction: a review. Body Image. 2008 Sep;5(3):244-50. doi: 10.1016/j.bodyim.2008.02.003. PMID 18424245
- [Background] Tiggemann M, Hayden S, Brown Z, Veldhuis J. The effect of Instagram "likes" on women's social comparison and body dissatisfaction. Body Image. 2018 Sep;26:90-97. doi: 10.1016/j.bodyim.2018.07.002. Epub 2018 Jul 21. PMID 30036748
- [Background] Leit RA, Gray JJ, Pope HG Jr. The media's representation of the ideal male body: a cause for muscle dysmorphia? Int J Eat Disord. 2002 Apr;31(3):334-8. doi: 10.1002/eat.10019. PMID 11920996
- [Background] Myers TA, Crowther JH. Social comparison as a predictor of body dissatisfaction: A meta-analytic review. J Abnorm Psychol. 2009 Nov;118(4):683-98. doi: 10.1037/a0016763. PMID 19899839
- [Background] Cahill S, Mussap AJ. Emotional reactions following exposure to idealized bodies predict unhealthy body change attitudes and behaviors in women and men. J Psychosom Res. 2007 Jun;62(6):631-9. doi: 10.1016/j.jpsychores.2006.11.001. PMID 17540220
- [Background] Arbour KP, Martin Ginis KA. Effects of exposure to muscular and hypermuscular media images on young men's muscularity dissatisfaction and body dissatisfaction. Body Image. 2006 Jun;3(2):153-61. doi: 10.1016/j.bodyim.2006.03.004. Epub 2006 May 19. PMID 18089218
- [Background] Fardouly J, Vartanian LR. Negative comparisons about one's appearance mediate the relationship between Facebook usage and body image concerns. Body Image. 2015 Jan;12:82-8. doi: 10.1016/j.bodyim.2014.10.004. Epub 2014 Nov 17. PMID 25462886
- [Background] Cafri G, Thompson JK, Ricciardelli L, McCabe M, Smolak L, Yesalis C. Pursuit of the muscular ideal: Physical and psychological consequences and putative risk factors. Clin Psychol Rev. 2005 Feb;25(2):215-39. doi: 10.1016/j.cpr.2004.09.003. Epub 2004 Dec 30. PMID 15642647
- [Background] Galioto R, Crowther JH. The effects of exposure to slender and muscular images on male body dissatisfaction. Body Image. 2013 Sep;10(4):566-73. doi: 10.1016/j.bodyim.2013.07.009. Epub 2013 Sep 3. PMID 24008185
- [Background] Tiggemann M, Zaccardo M. "Exercise to be fit, not skinny": The effect of fitspiration imagery on women's body image. Body Image. 2015 Sep;15:61-7. doi: 10.1016/j.bodyim.2015.06.003. Epub 2015 Jul 10. PMID 26176993